CLINICAL TRIAL: NCT04789330
Title: The Choice of Vasopressor for Treating Hypotension During General Anesthesia: a Pilot Pragmatic Cluster Cross-over Randomized Trial (the VEGA-1 Trial)
Brief Title: Norepinephrine vs Phenylephrine During General Anesthesia
Acronym: VEGA-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: A135759
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Surgery; Hypotension
Keywords: vasopressor; outcome; AKI; cardiovascular; complications
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Intervention Model Description: pragmatic, cluster-randomized, open-labeled, multiple-crossover trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Norepinephrine (Active Comparator): Norepinephrine continuous infusion as the first line vasopressor
  Interventions: Drug: Norepinephrine
- Phenylephrine (Active Comparator): Phenylephrine continuous infusion as the first line vasopressor
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine administered during anesthesia
  Arms: Norepinephrine
Drug: Phenylephrine — Phenylephrine administered during anesthesia
  Arms: Phenylephrine

SUMMARY:
50 million patients undergo surgery each year in the United States. Postoperative mortality is considered the third leading cause of death worldwide. Hypotension during surgery have been linked to increased postoperative morbidity and mortality. Episodes of hypotension during surgery are associated with an increased risk of acute kidney injury, stroke, cardiac events and death. Treating or preventing hypotension during general anesthesia and major surgery was found to improve outcomes. At this time, it is unclear what is the best vasopressor to maintain blood pressure during surgery under general anesthesia. With this pilot pragmatic trial, the investigators will explore the impact of norepinephrine (NE) or phenylephrine (PE) on post-operative events in patients undergoing major surgery with general anesthesia and needing vasopressors infusion to maintain their systemic arterial pressure.

DETAILED DESCRIPTION:
Postoperative mortality is considered the third leading cause of death worldwide. Hemodynamic instability and specifically hypotension during surgery have been linked to increased postoperative morbidity and mortality. Episodes of hypotension during surgery are associated with an increased risk of acute kidney injury, stroke, cardiac events and death. Treating or preventing hypotension during general anesthesia and major surgery was found to improve outcomes. At this time, it is unclear what is the best vasopressor to maintain blood pressure during surgery.

Hypotension during anesthesia and surgery is commonly treated with vasopressors such as phenylephrine (PE), a synthetic pure vasoconstrictor, or norepinephrine (NE), which has both inotropic and vasoconstrictor activity. NE increases cardiac output and increases cardio-vascular coupling due to alpha-agonist effects compared to PE, a purely vasoconstrictive agent.

The investigators hypothesize that norepinephrine will be superior to phenylephrine. The effect size is expected to be modest, therefore requiring a large sample size, and will vary between subgroups determined by patients' individual characteristics.

This pilot trial (VEGA-1) will allow to 1) test the feasibility of the study using a cross-over cluster randomized controlled trial and 2) estimate the effect size of the use of NE or PE on post-operative outcome in the overall population but also investigate the Heterogeneity in Treatment Effect (HTE) of the drugs among subgroups or clusters of patients for designing a larger trial.

Design: pragmatic, cluster-randomized, open-labeled, multiple-crossover trial across hospital from University of California, San Francisco (UCSF) and University of California, Los Angeles (UCLA). Centers will be assigned to use either PE or NE for the first-line intravenous infusion of vasopressor in the OR. Data will be collected in routine clinical care and automatically extracted from the electronic health record (EHR).

Primary endpoint:

- Separation between study groups in the first line vasopressor administration (% of cases with appropriate vasopressor with respect to group attribution).

Secondary endpoints:

* Death within 30 days
* Acute kidney injury defined by the KDIGO definition
* Severe acute kidney injury (stage 2 or 3 of the KDIGO definition)
* Myocardial Injury following non-cardiac surgery (MINS)
* Adverse cardio-renal events
* Hospital length of stay
* Rehospitalization within 30 days

ELIGIBILITY:
Inclusion Criteria:

* age 18 Years and older
* Surgery under general anesthesia and requiring infusion of vasopressors to maintain the mean arterial pressure.
* Surgery duration>2 hours

Exclusion Criteria:

* Cardiac surgery
* Patients on ECMO
* Organ transplantation
* Outpatient (come-and-go surgery)
* Obstetric procedures
* Patient already receiving NE or PE before induction of anesthesia
* Patients transferred immediately (i.e. within 24 hours) after surgery to another hospital.
* Patients with severe trauma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3626 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu LEGRAND, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center at Mount Zion, San Francisco, California
  - UCSF Medical Center at Parnassus, San Francisco, California
  - UCSF Medical Center at Mission Bay, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Legrand M, Kothari R, Fong N, Palaniappa N, Boldt D, Chen LL, Kurien P, Gabel E, Sturgess-DaPrato J, Harhay MO, Pirracchio R, Bokoch MP; VEGA-1 trial investigators. Norepinephrine versus phenylephrine for treating hypotension during general anaesthesia in adult patients undergoing major noncardiac surgery: a multicentre, open-label, cluster-randomised, crossover, feasibility, and pilot trial. Br J Anaesth. 2023 May;130(5):519-527. doi: 10.1016/j.bja.2023.02.004. Epub 2023 Mar 14. PMID 36925330
- [Derived] Krone S, Bokoch MP, Kothari R, Fong N, Tallarico RT, Sturgess-DaPrato J, Pirracchio R, Zarbock A, Legrand M. Association between peripheral perfusion index and postoperative acute kidney injury in major noncardiac surgery patients receiving continuous vasopressors: a post hoc exploratory analysis of the VEGA-1 trial. Br J Anaesth. 2024 Apr;132(4):685-694. doi: 10.1016/j.bja.2023.11.054. Epub 2024 Jan 19. PMID 38242802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Over a 6-month period, participating sites were randomized to an alternating sequence of first-line vasopressor use. Three sites were randomized to start with Norepinephrine (NE), and two clinics were randomized to start with Phenylephrine (PE). All five sites used each vasopressor (NE and PE) for 3 months.
Pre-assignment Details: To maintain a de-identified dataset, the date of participant enrollment/surgery was not collected. Therefore. the Participant Flow cannot be presented according to the sequence assigned to the sites, as the number of participants enrolled in each site per month was not collected, nor can it be derived. Data are reported according to the total number of participants randomized to NE and PE and sites are not shown as the units assigned to avoid double-counting sites in the Participant Flow.
Groups:
- Norepinephrine: Continous infusion of Norepinephrine as the first-line vasopressor during anesthesia
- Phenylephrine: Continuous infusion of phenylephrine as the first-line vasopressor during anesthesia
Period: Overall Study
Arm/Group | Norepinephrine | Phenylephrine
Started | 1809 | 1817
Site 1 (Randomized to NE first, then PE, then NE, then PE, then NE, then PE months 1-6) | 845 | 815
Site 2 (Randomized to PE first, then NE, then PE, then NE, then PE, Then NE months 1-6) | 302 | 310
Site 3 | 110 | 128
Site 4 | 261 | 289
Site 5 | 291 | 275
Completed | 1809 | 1817
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Norepinephrine: Norepinephrine continuous infusion as the first-line vasopressor
- Phenylephrine: Phenylephrine continuous infusion as the first-line vasopressor
- Total: Total of all reporting groups
Arm/Group | Norepinephrine | Phenylephrine | Total
Number analyzed (Participants) | 1809 | 1817 | 3626
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [50 to 72] | 63 [50 to 72] | 63 [50 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 917 | 908 | 1825
  Male | 892 | 909 | 1801
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 326 | 308 | 634
  Not Hispanic or Latino | 1440 | 1469 | 2909
  Unknown or Not Reported | 43 | 40 | 83
Region of Enrollment [Number; unit: participants]
  United States | 1809 | 1817 | 3626

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Assigned Vasopressor Given
Description: First line vasopressor administration will be measured as a percent of total eligible participants with assigned vasopressor given during anesthesia time, up to 24 hours
Time Frame: Anesthesia time, up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Norepinephrine | Phenylephrine
Number analyzed (Participants) | 1809 | 1817
Participants | 1570 | 1627

2. Secondary Outcome: Number of Participants Who Died Within 30 Days After Surgery
Description: Death within 30 days of surgery.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Norepinephrine | Phenylephrine
Number analyzed (Participants) | 1809 | 1817
Participants | 20 | 22

3. Secondary Outcome: Number of Participants With Acute Kidney Injury (AKI)
Description: AKI is measured using the Kidney Disease: Improving Global Outcomes (KDIGO) definition based on serum creatinine. Acute kidney injury is defined as an increase in serum creatinine ≥ 0.3 mg/dL within 48 hours, or an increase in serum creatinine ≥ 1.5-fold from baseline within 7 days, or initiation of renal replacement therapy within 7 days.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Norepinephrine | Phenylephrine
Number analyzed (Participants) | 1809 | 1817
Participants | 140 | 135

4. Secondary Outcome: Number of Participants With Severe Acute Kidney Injury
Description: Severe acute kidney injury is assessed using the KDIGO definition based on serum creatinine or need for Renal Replacement Therapy (RRT). Severe Acute Kidney Injury is defined as an increase in serum creatinine ≥ 2-fold from baseline within 7 days, or initiation of renal replacement therapy within 7 days.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Norepinephrine | Phenylephrine
Number analyzed (Participants) | 1809 | 1817
Participants | 28 | 31

5. Secondary Outcome: Hospital Length of Stay
Description: Days between date of surgery and hospital discharge
Time Frame: In-hospital, up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Norepinephrine | Phenylephrine
Number analyzed (Participants) | 1809 | 1817
days | 4 [2.1 to 7.0] | 4.1 [2.1 to 7.5]

6. Secondary Outcome: Number of Participants With Myocardial Injury After Non-cardiac Surgery (MINS)
Description: Number of participants with post-operative myocardial injury defined as a troponin elevation.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Norepinephrine | Phenylephrine
Number analyzed (Participants) | 1809 | 1817
Participants | 44 | 38

7. Secondary Outcome: Adverse Cardio-renal Events
Description: Number of patients meeting a combined endpoint of AKI and/or MINS
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Norepinephrine | Phenylephrine
Number analyzed (Participants) | 1809 | 1817
Participants | 168 | 159

8. Secondary Outcome: Rehospitalization Within 30 Days
Description: Patients discharge and readmitted for more than 24 hours within 30 days after surgery
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Norepinephrine | Phenylephrine
Number analyzed (Participants) | 1809 | 1817
Participants | 56 | 66

ADVERSE EVENTS:
Time Frame: Mortality was collected until 30 days post-surgery, and other adverse events were collected until 7 days post-surgery.
Arm/Group | Norepinephrine | Phenylephrine
All-Cause Mortality (participants affected / at risk) | 20/1809 | 22/1817
Serious Adverse Events (participants affected / at risk) | 20/1809 | 22/1817
Other Adverse Events (participants affected / at risk) | 168/1809 | 159/1817
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norepinephrine (N=1809) | Phenylephrine (N=1817)
mortality (Cardiac disorders) | 20 (20) | 22 (22)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norepinephrine (N=1809) | Phenylephrine (N=1817)
Acute Kidney Injury (Renal and urinary disorders) | 140 (140) | 135 (135) — Occurrence of AKI within 7 days of surgery.
Myocardial injury (Cardiac disorders) | 44 (44) | 38 (38) — Myocardial injury, troponin greater than 99th percentile of normal within 7 days of surgery.

LIMITATIONS AND CAVEATS:
Pragmatic trial with events recorded throughout the eHR

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT04789330/Prot_SAP_000.pdf